CLINICAL TRIAL: NCT00679549
Title: The Role of Sleep Apnea in the Acute Exacerbation of Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Rami Khayat, Associate Professor-Clinical, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008H0011
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Results first posted 2019-05-14 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-04

CONDITIONS: Heart Failure; Obstructive Sleep Apnea; Heart Failure, Congestive
Keywords: Heart Failure; Obstructive Sleep Apnea; OSA; CHF; Sleep apnea; CHD
MeSH Terms: conditions — Heart Failure; Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DEVICE (Experimental): Provided CPAP as an inpatient
  Interventions: Device: CPAP Therapy
- Control (No Intervention): No device provided

INTERVENTIONS:
Device: CPAP Therapy — CPAP therapy is provided as an inpatient.
  Other Names: CPAP Device
  Arms: DEVICE

SUMMARY:
This study will evaluate whether treating sleep apnea while in the hospital would help heart failure, and assist recovery from the worsening of the heart function more than the current clinical standard of waiting for treatment until the subject have left the hospital.

Heart failure affects more than 2% of the US population and is the only cardiovascular disorder with rising incidence. The annual cost of CHF in 2005 was $ 27.9 billion, large percentage of which is the cost of hospitalizations for exacerbation of CHF. Half of patients with CHF have some form of sleep apnea, and most of them go undiagnosed. Patients with CHF and OSA benefit from treatment with CPAP as an outpatient. The society can benefit from developing recommendations for approaching sleep apnea in the hospitalized CHF patient, which may shorten length of stay, improve functional status of discharged patient, and reduce rehospitalizations.

DETAILED DESCRIPTION:
Target population:

Patients admitted to the OSU Heart Hospital with ADHF routinely undergo a cardiorespiratory sleep study to identify OSA. Patients with ADHF who are newly diagnosed with OSA during the same hospital stay are eligible for this study.

Enrollment:

Given the presence of significant previously unrecognized OSA in 62% of patients hospitalized with ADHF, we expect to need to screen 270 patient volunteers to recruit 170 patients with OSA.

Eligibility for randomization: The criteria for ADHF is admission diagnosis of heart failure; a chief complaint of dyspnea; and ejection fraction of 45% or less. Additionally, elevated left ventricular pressure as indicated by at least one sign and one symptom of volume overload (pedal edema, crackles, consistent chest X-ray, increased left ventricular end-diastolic diameter, or elevated BNP level) is required [46].

ELIGIBILITY:
Inclusion Criteria:

* Previously unrecognized OSA with an Apnea Hypopnea Index (AHI) > 15 events per hour on the attended in-hospital sleep study. Patients with apnea index of less than 5 events / hour are excluded (see design consideration for rationale)
* Projected length of stay 3 days or more on the morning following the cardio-respiratory sleep study
* Ongoing or planned targeted treatment for heart failure including one of the following: IV diuretics, IV infusion of inotropes or vasodilators, or planned revascularization, or device therapy

Exclusion Criteria:

* Patients who are already diagnosed with OSA
* Patients with Central Sleep Apnea
* Patients with diastolic only heart failure
* Cardiogenic shock and hemodynamic instability with MAP less than 55 mmHg off vasopressors, or concurrently on vasopressor treatment, left ventricular assist devices, or intra-aortic Balloon Pump. Inotropic agents will not constitute an exclusion criterion. Patients will be eligible once off vasopressors.
* Acute respiratory failure or insufficiency defined by P/F (PaO2/FIO2) ratio less than 250, or FIO2 requirement more than 50%
* Overt neurological deficit
* Renal failure requiring renal replacement therapy; Patients will not be excluded if they were undergoing ultra-filtration for volume removal
* Patients scheduled for procedures that will interfere with post randomization measurement: This includes scheduled coronary bypass surgery, or expected left ventricular assist device placement.
* Patients who arrived from a long-term care facility or expected to be discharged to one; and patients who have very poor functional outcome precluding ability to use the CPAP device independently.
* Patients on long term or "bridging" inotropic infusion, or short life expectancy due to concomitant illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2008-03; Primary Completion 2014-03-22 (Actual); Study Completion 2014-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rami N Khayat, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 150 patients provided the baseline measurements and were randomized and included in the trial.
Period: Overall Study
Arm/Group | DEVICE | Control
Started | 75 | 75
Completed | 69 | 66 (4 dropouts in the control arm; 5 missing echocardiograms in the control arm)
Not Completed | 6 | 9
Not completed — dropout | 2 | 4
Not completed — missing outcome echocardiograms | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DEVICE | Control | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (11) | 57 (13.5) | 57 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 21 | 43
  Male | 53 | 54 | 107
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 18 | 17 | 35
  White | 57 | 58 | 115

OUTCOME MEASURES:

1. Primary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: Using the modified Simpson method. LVEF is calculated as (Left ventricular end diastolic volume (LVEDV)-left ventricular end systolic volume (LVESV)/left ventricular end diastolic volume (LVEDV) *100.
  the measurement unit of LVEF is %.
Time Frame: at baseline and 3 days post randomization
Measure: Mean (Standard Deviation); unit: percent ejection fraction
Arm/Group | DEVICE | Control
Number analyzed (Participants) | 69 | 66
percent ejection fraction
  Baseline | 25.3 (10.6) | 27.0 (11.3)
  Conclusion | 27.3 (11.9) | 28.8 (10.5)

ADVERSE EVENTS:
Time Frame: 3 months post randomization
Arm/Group | DEVICE | Control
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/75
Other Adverse Events (participants affected / at risk) | 0/75 | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No